CLINICAL TRIAL: NCT00744640
Title: Gemcitabine, Oxaliplatin and Capecitabine (GEMOXEL) for Patients With Advanced Pancreatic Adenocarcinoma (APC): A Phase I/II Study
Brief Title: Gemcitabine, Oxaliplatin and Capecitabine for Advanced Pancreatic Carcinoma
Acronym: GEMOXEL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Cancer League (Other); Roche Pharma AG (Industry); Sanofi (Industry)
Responsible Party: Dr. Viviane Hess, University Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK-Nr. 92/05; 2005DR2296
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Locally Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: advanced pancreatic cancer; palliative chemotherapy; first-line therapy; capecitabine; oxaliplatin; gemcitabine; dose-finding study; Phase II
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): single arm study with triple combination chemotherapy
  Interventions: Drug: gemcitabine, oxaliplatin, capecitabine

INTERVENTIONS:
Drug: gemcitabine, oxaliplatin, capecitabine — gemcitabine day 1 and 8, oxaliplatin day 1, capecitabine days 1-14, q3weeks

SUMMARY:
Gemcitabine is the mainstay of palliative chemotherapy for patients with advanced pancreatic cancer (APC). Recent randomized trials have shown increased clinical benefit with the addition of oxaliplatin and prolonged median survival with the addition of capecitabine to gemcitabine. Gemcitabine, capecitabine and oxaliplatin are 3 newer, well tolerated anticancer drugs with mild and non-overlapping toxicity profiles. We therefore propose a dose-finding and safety study of the triple combination gemcitabine, capecitabine and oxaliplatin in patients with APC (Phase I part), followed by a phase II part to assess preliminary efficacy of this triple combination.

DETAILED DESCRIPTION:
Primary Objectives:

* Phase I: to determine the maximum tolerated dose (MTD) of oxaliplatin in combination with gemcitabine and capecitabine (GEMOXEL) in patients with APC
* Phase II: to assess any anti-tumor activity of GEMOXEL in patients with APC

Secondary Objectives:

* to assess toxicity and safety of the combination treatment GEMOXEL in patients with APC

Primary Endpoints:

* Phase I: Dose-limiting toxicity
* Phase II: Objective tumor response

Secondary Endpoints:

* Toxicity at MTD according to NCI CTC 3.0
* Progression-free survival and Overall Survival

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed adenocarcinoma of the exocrine pancreas
* Disease non-resectable and locally advanced or metastatic
* Measurable disease or evaluable disease i.e. tumor marker CA19-9 at baseline ≥ 1.5 x upper limit of normal (ULN)
* Age >18 years
* Karnofsky performance status ≥ 60%
* Life expectancy of at least 3 months
* Written informed consent
* Willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Prior chemotherapy for pancreatic cancer
* Prior adjuvant radio- or radiochemotherapy for pancreatic cancer within 12 months of inclusion
* Known CNS metastases at the time of enrollment
* Neutrophil count ≤ 1.5 x109/l, platelet count ≤100 x109/l, hemoglobin ≤ 10g/dl
* Serum creatinine > 1.25 x ULN
* ASAT, ALAT and alkaline phosphatase > 2.5 ULN or > 5 ULN in the presence of liver metastasis, Bilirubin > 1.5 ULN (after treatment of obstructive jaundice eg. stent)
* Pregnant or breast feeding women (women of childbearing potential must have a negative pregnancy test at baseline)
* Men and women of reproductive potential who are not using an effective method of contraception
* Clinically significant cardiac disease (NYHA III-IV) or myocardial infarction within the last 12 months
* Neurological disease with dys-/paraesthesias > grade 1 according to NCI CTC
* Any serious concomitant disorder incompatible with the trial (in the judgement of the investigator)
* Psychiatric disability thought to be clinically significant in the opinion of the investigator precluding informed consent or interfering with compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 weeks

SECONDARY OUTCOMES:
Progression-free survival and overall survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Hess, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (8):
- Switzerland (8):
  - Cantonal Hospital Bruderholz, Bruderholz, Basel-Landschaft
  - Cantonal Hospital Liestal, Liestal, Basel-Landschaft
  - St. Clara Hospital, Basel
  - University Hospital Basel, Basel
  - Cantonal Hospital Lucerne, Lucerne
  - City Hospital Triemli, Zurich
  - Oncocenter Hirslanden, Zurich
  - University Hospital, Zurich